CLINICAL TRIAL: NCT05002725
Title: A Comparison of Quadriceps Muscle Weakness Associated With PENG Blockade or Femoral Nerve Blockade for Patients Undergoing Neck of Femur (NOF) Fracture Surgery
Brief Title: PENG Versus Femoral Nerve Block in Neck of Femur Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Collaborators: Health Service Executive (Unknown)
Responsible Party: Principal Investigator, Brian Declan O'Donnell, Clinical Senior Lecturer, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCCork 2021-BOD-1
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Neck of Femur Fracture
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This will be a double blinded study where patients and assessors are blinded to the technique used. The operator performing the block cannot be blinded. It will not be possible to tell from the appearance of the catheter whether it is a femoral nerve catheter or PENG catheter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG (Experimental): An ultrasound guided PENG catheter will be inserted. 20ml of 1.5% lidocaine will be administered.
  Interventions: Drug: Lidocain
- Femoral Block (Active Comparator): An ultrasound guided Femoral Nerve catheter will be inserted. 20ml of 1.5% lidocaine will be administered.
  Interventions: Drug: Lidocain

INTERVENTIONS:
Drug: Lidocain — 300mg (20ml) will be injected

SUMMARY:
Neck of femur (NOF) fracture is a common presentation to the emergency department, particularly in our older population. NOF fracture is associated with a high social and economic cost with significant effects on patients' quality of life. Analgesia and ambulation are important determinants of outcome following NOF surgery. We propose to compare whether PENG or Femoral Nerve Block is associated with a greater degree of quadriceps motor dysfunction.

DETAILED DESCRIPTION:
Neck of femur (NOF) fracture is a common presentation to the emergency department, particularly in our older population.1.NOF fracture is associated with a high social and economic cost with significant effects on patients' quality of life

The latest Irish Hip Fracture Database (IHFD) report from 2019 detailed 3,701 NOF fractures in patients over 60 years of age in Ireland and 437 of these patients attended CUH.2 This frail and vulnerable group had an average age of 81 and many people suffered numerous co-morbid conditions. 3 This population of patients is therefore at significant risk of complications and require multidisciplinary input to optimise clinical outcome

From a patient's perspective, NOF fracture is a very painful condition, requiring early surgical fixation. It is associated with significant morbidity and mortality. In 2019, 5% of patients who sustained a hip fracture in Ireland died, an additional 4% of patients required new admission to a nursing home following this fracture and a further 13% required convalescent care3

These patients are also particularly at risk for under-treatment of pain. Contraindications to many commonly used analgesics such as non-steroidal anti-inflammatory drugs (NSAIDs) exist in this population, including renal dysfunction in 40%5. Older adults suffer more adverse effects from opiate analgesia such as nausea, vomiting, constipation, drowsiness and respiratory complications. This population also have a 25% incidence of cognitive impairment which may make communication and assessment of their pain more challenging. 1, 3 Under-treated pain also confers a 9 fold increased risk of delirium in cognitively intact patients14

Peripheral nerve blocks (PNB) have been extensively researched in this group of patients with a view to improving the quality of pain relief while reducing the side effects of analgesic medications used. In 2017, a Cochrane review on PNB in the management of patients with NOF fractures concluded that there was high quality evidence that PNB reduces pain on movement within 30 minutes after block placement and reduces opioid consumption and moderate quality evidence that PNB reduces the incidence of pneumonia, time to first mobilization and cost. 6

Widespread use of PNB on admission to hospital and in the early postoperative period is also supported by the latest Association of Anaesthetists' (AoA) guideline: "Guideline for the management of hip fractures 2020". In this, they recommend using femoral or fascia iliaca blocks as pericapsular nerve group (PENG) blocks have not yet been compared with these more established blocks in trials. They also recommend that general anaesthesia or spinal anaesthesia should be routinely supplemented with PNB and state that there is little evidence at present for continuous catheter techniques which may delay remobilisation5

Issues with current practice:

Often patients with NOF fractures endure significant pain during their hospitalisation. The proportion of patients receiving PNB varies nationally from 10-95% depending on hospital. The AoA recommend that PNB should be undertaken in the Emergency department and at the time of surgery provided 6 hours have passed.5 Under-treated pain has been demonstrated to increase the risk of delirium in cognitively intact patients with NOF fractures with a relative risk of 9.014 It is also likely to lead to significant patient dissatisfaction Single injection PNB blocks are limited by short duration a fact that can be mitigated by continuous catheter techniques. A study from our institution published in 2012 demonstrated more effective perioperative analgesia, reduced opiate consumption and improved patient satisfaction when continuous femoral nerve blockade was compared with a standard opiate based regime in patients with NOF fractures.7 However, femoral nerve blockade can be associated with weakness of the quadriceps muscle, possibly reducing early postoperative mobility and increasing the risk of falls. A study of healthy volunteers demonstrated a significant reduction in quadriceps strength and balance scores following femoral nerve blockade8 Another study suggested a causal relationship between continuous peripheral nerve blocks and falls after hip and knee arthroplasty 9

Proposal of novel intervention We propose performing a PENG block for postoperative analgesia. The pericapsular nerve group (PENG) block, first described in 2018, is a PNB technique which aims to provide analgesia for patients with NOF fractures by blocking sensory branches of the femoral nerve, obturator nerve and accessory obturator nerve to the anterior hip capsule.10

Justification in support of the intervention The PENG block aims to block the articular branches of the femoral, obturator and accessory obturator nerves which supply the hip joint.10 Tran et al demonstrated spread to all three nerves using the PENG block technique.11This is theoretically a more comprehensive blockade of the pain fibres from the hip than would be achieved with a traditional femoral nerve block. Therefore the analgesia achieved may be superior than with other blocks. Published case reports and case series suggest PENG block efficacy.13

The PENG block aims to block the sensory articular branches while sparing the motor innervation of the quadriceps muscle. This is likely to result in less quadriceps muscle weakness which in turn can affect balance and may cause contribute to falls postoperatively.8,9

The AoA do not recommend continuous catheter techniques in their latest guideline due to a lack of evidence and the potential contribution of quadriceps weakness to falls.5 If the PENG block does not cause quadriceps weakness and has the potential to provide superior analgesia, this is likely to improve a patient's ability to mobilise early postoperatively and engage with physiotherapy and rehabilitation. This may improve outcomes. Continuous catheter techniques (most commonly PENG catheters) are currently used in our institution for postoperative analgesia

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for operative repair of hip fracture Patient age 16 years or more ASA I - III

Exclusion Criteria:

* Patient refusal Coagulopathy Local infection Allergy to Local Anaesthetics Significant cognitive impairment (4AT score>=4) Weight <60kg

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Quadriceps Motor Block | 20 mins post procedure
  Presence or absence of motor block

SECONDARY OUTCOMES:
Pain | 20 mins post procedure
  VRS on passive hip flexion
12 hr Pain | 20 mins post procedure
  VRS on passive hip flexion
24 hr Pain | 20 mins post procedure
  VRS on passive hip flexion
Quadriceps Motor block | 24 hours post op
  Present or absent
cumulative opiate consumption | 24 hours post op

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided